CLINICAL TRIAL: NCT01268358
Title: A Single Center, Open-label, Dose Escalation Study of the Safety and Pharmacokinetics of rhLAMAN (Recombinant Human Alpha-mannosidase or Lamazym) for the Treatment of Patients With Alpha-mannosidosis.
Brief Title: Safety Study of Recombinant Human Alpha-mannosidase for the Treatment of Patients With Alpha-mannosidosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zymenex A/S (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rhLAMAN-02; 2010-022084-36 (EudraCT Number)
Record Dates: First submitted 2010-12-29; First posted 2010-12-30 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Alpha Mannosidosis
MeSH Terms: conditions — alpha-Mannosidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Lamazym 6.25 (Experimental)
  Interventions: Drug: Lamazym
- Lamazym 12.5 (Experimental)
  Interventions: Drug: Lamazym
- Lamazym 25 (Experimental)
  Interventions: Drug: Lamazym
- Lamazym 50 (Experimental)
  Interventions: Drug: Lamazym
- Lamazym 100 (Experimental)
  Interventions: Drug: Lamazym

INTERVENTIONS:
Drug: Lamazym — Lamazym, ERT, infusion weekly
  Other Names: rhLAMAN

SUMMARY:
This is a single-center, open-label, dose escalation study of patients with alpha-mannosidosis. 10 patients will be enrolled in this study receiving intravenous infusions of Lamazym. In order to avoid development of delayed hypersensitivity all patients will continue weekly treatment at the designated dose until the Safety Committee approves transfer to the rhLAMAN-03 protocol.

It is the hypothesis that Lamazym is safe to use.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have a confirmed diagnosis of alpha-mannosidosis as defined by alpha-mannosidase activity < 10% of normal activity in blood leukocytes
2. The patient must have an age at the time of screening ≥ 5 year and ≤ 20 years
3. The patient must have physical ability to perform 6-minutes walk test (6MWT), 3 minute-stair climb test (3MSCT) and pulmonary lung function test (spirometry, body plethysmography).
4. The patient must have the ability to mentally cooperate in the cognitive and motor function tests
5. The patient must have the ability to hear and follow a request. Hearing aids can be worn.
6. Patient or patient's legally authorized guardian(s) must provide signed, informed consent prior to performing any study-related activities (trial-related activities are any procedures that would not have been performed during normal management of the subject)
7. The patient and his/her guardian(s) must have the ability to comply with the protocol

Exclusion Criteria:

1. The patient cannot walk without support.
2. Presence of known chromosomal abnormality and syndromes affecting psychomotor development, other than alpha-mannosidosis
3. History of bone marrow transplantation
4. Presence of known clinically significant cardiovascular, hepatic, pulmonary or renal disease or other medical conditions that, in the opinion of the Investigator, would preclude participation in the trial
5. Presence of an ECHO with abnormalities within half a year that, in the opinion of the Investigator, would preclude participation in the trial
6. Any other medical condition or serious intercurrent illness, or extenuating circumstance that, in the opinion of the investigator, would preclude participation in the trial
7. Pregnancy
8. Psychosis within the last 3 months

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety profile of rhLAMAN (Lamazym) | 1-5 weeks

SECONDARY OUTCOMES:
To determine the PK profile of rhLAMAN (Lamazym) in patients with alpha-mannosidosis as measured by rhLAMAN levels in plasma | 1 dosis
To collect baseline measurements that are to be used for efficacy evaluation in the following trial (rhLAMAN-03) | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Allan M. Lund, MD, Principal Investigator — Department of Clinical Genetics, Juliane Marie Centre, Region Hovedstaden, Copenhagen University hospital, Denmark; Jens Fogh, Study Chair — Zymenex A/S

REFERENCES:
- [Background] Borgwardt L, Thuesen AM, Olsen KJ, Fogh J, Dali CI, Lund AM. Cognitive profile and activities of daily living: 35 patients with alpha-mannosidosis. J Inherit Metab Dis. 2015 Nov;38(6):1119-27. doi: 10.1007/s10545-015-9862-4. Epub 2015 May 28. PMID 26016802
- [Result] Borgwardt L, Dali CI, Fogh J, Mansson JE, Olsen KJ, Beck HC, Nielsen KG, Nielsen LH, Olsen SO, Riise Stensland HM, Nilssen O, Wibrand F, Thuesen AM, Pearl T, Haugsted U, Saftig P, Blanz J, Jones SA, Tylki-Szymanska A, Guffon-Fouiloux N, Beck M, Lund AM. Enzyme replacement therapy for alpha-mannosidosis: 12 months follow-up of a single centre, randomised, multiple dose study. J Inherit Metab Dis. 2013 Nov;36(6):1015-24. doi: 10.1007/s10545-013-9595-1. Epub 2013 Mar 14. PMID 23494656
- [Result] Borgwardt L, Stensland HM, Olsen KJ, Wibrand F, Klenow HB, Beck M, Amraoui Y, Arash L, Fogh J, Nilssen O, Dali CI, Lund AM. Alpha-mannosidosis: correlation between phenotype, genotype and mutant MAN2B1 subcellular localisation. Orphanet J Rare Dis. 2015 Jun 6;10:70. doi: 10.1186/s13023-015-0286-x. PMID 26048034
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2010-022084-36